CLINICAL TRIAL: NCT04635995
Title: An Open Label, First in Human (FIH), Phase 1a/1b Trial of LVGN7409 (CD40 Agonist Antibody) as a Single Agent, in Combination With LVGN3616 (Anti-PD-1 Antibody), and in Combination With LVGN3616 and LVGN6051 (CD137 Agonist Antibody) in Patients With Locally Advanced, Relapsed, Refractory, or Metastatic Malignancy
Brief Title: Phase 1 Trial of LVGN7409 (CD40 Agonist Antibody) as Single Agent and Combination Therapies in Advanced or Metastatic Malignancy
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Lyvgen Biopharma Holdings Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LVGN7409-101
Record Dates: First submitted 2020-11-09; First posted 2020-11-19 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Cancer
Keywords: Lyvgen; CD40
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Monotherapy dose escalation (Experimental): The monotherapy dose escalation phase includes 8 dose levels of LVGN7409. Route of administration is IV infusion, and the frequency of administration is once every 3 weeks (Q3W). One cycle is 3 weeks, and treatment can be up to 35 cycles if patients receive benefits.
  Interventions: Biological: LVGN7409

INTERVENTIONS:
Biological: LVGN7409 — IV infusion once every 3 weeks (Q3W).

SUMMARY:
LVGN7409 is a humanized monoclonal antibody that specifically binds to CD40, and acts as an agonist against CD40.

This first in human study of LVGN7409 is designed to establish the maximum tolerated dose (MTD) and/or the recommended dose for expansion (RDE) as well as the recommended Phase 2 dose(s) (RP2D) of LVGN7409, both as a single agent (monotherapy) and in combination with a fixed dose of anti-PD-1 antibody and/or CD137 agonist in the treatment of advanced or metastatic malignancy.

DETAILED DESCRIPTION:
This is an open-label, non-randomized, two-stage, FIH Phase 1 study, utilizing an accelerated dose escalation followed by a traditional 3 + 3 dose escalation algorithm to identify the MTD and/or RDE and RP2D of LVGN7409 as a single agent (monotherapy) and in combination with anti-PD-1 antibody and/or CD137 agonist. The first stage of the study is the dose escalation phase (i.e., Phase 1a). The second stage of the study is the dose expansion phase (i.e., Phase 1b). During the study, dose interruption(s) and/or delay(s) may be implemented based on toxicity. Dose modifications are not permitted. Intra-patient dose escalations will be allowed for the early dose cohorts (single-patient dose groups) in Phase 1a Part 1. Patients will be considered evaluable for safety and tolerability if they receive at least one dose of LVGN7409 or anti-PD-1 antibody and/or CD137 agonist at the specified cohort dose. Patients in all parts of the trial will remain on therapy until confirmed disease progression or for 2 years, whichever occurs first. However, patients who are clinically unstable will discontinue following the initial assessment of disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged ≥ 18 years.
* Ability to understand and willingness to sign a written informed consent document.
* Patients must have a histologically or cytologically confirmed metastatic or unresectable malignancy.
* Estimated life expectancy, in the judgment of the Investigator, of at least 90 days.
* Adequate bone marrow, liver, and renal functions
* Men and women of childbearing potential must agree to take highly effective contraceptive methods.
* Patients should recover from all reversible AEs of previous anticancer therapies to baseline.
* Patients infected with the HIV virus will be eligible if the disease is under control of effective therapy.

Exclusion Criteria:

* Prior therapy with anti-CD40 therapy.
* Receipt of systemic anticancer therapy or radiotherapy within certain period of time.
* Prior exposure to immune-therapeutics experienced Grade ≥ 3 drug-related toxicity, or a toxicity requiring discontinuation.
* Received a live-virus vaccine within 30 days of the first dose of study drug.
* Grade ≥ 3 allergic reaction to treatment with a monoclonal antibody.
* History of Grade ≥ 3 immune-related AEs (irAEs).
* Prolonged QT syndrome, or clinically significant cardiac condition.
* Receiving an immunologically based treatment for any reason.
* History or current active or chronic autoimmune disease.
* Uncontrolled pleural effusion, pericardial effusion, or recurrent ascites drainage.
* Female patients who are pregnant or breastfeeding.
* History of hemorrhagic or ischemic stroke within the last 6 months.
* Previously received an allogeneic tissue/organ transplant, stem cell or bone marrow transplant or solid organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2020-12-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Treatment-emergent adverse events (TEAEs) | up to 24 months
  determination of DLTs and serious AEs (SAEs) of LVGN7409 as monotherapy. Adverse events will be assessed, and severity will be assigned by using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0
RP2D of LVGN7409 as monotherapy | up to 24 months
  determination of MTD, RDE and/or RP2D of LVGN7409 as monotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States